CLINICAL TRIAL: NCT06320119
Title: Setting a PERSONalized Outcome in ASthma: the PERSONAS Study. A Patient Driven Outcome (PDO) Study
Acronym: PERSONAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2943
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personal approach on asthma control (PDO group) (Experimental)
  Interventions: Other: PDO Group
- Non-personalized approach (UC group) (No Intervention)

INTERVENTIONS:
Other: PDO Group — Patients in the intervention gruop with set a personalized outcome within a usual asthma review consultation
  Arms: Personal approach on asthma control (PDO group)

SUMMARY:
To optimize the effectiveness of asthma therapy there is a need to identify and address individual patient goals. Considering the self-management discussion as central for the achievement of health outcomes, Healthcare Providers may help patients make specific actions to obtain their desired goals.

The current evidence suggest that Healthcare Professionals need to develop a more patient-centered and partnership-based approach based on the development and review of action plans, including the experiential asthma knowledge of patients and caregivers. From a practical perspective, the specialist (i.e. pulmunologists, allergologists, etc) has clear therapeutic targets to be reached in asthmatic patients: for example, improving the disease control, the spirometric values and asthma control test (ACT) score vs. pre-treatment evaluations represent the standard outcomes to reach (GINA 2019). However, as previously described, patients are more likely to achieve an improved clinical outcome when the treatment is driven by a personalized goal. This builds on the same principle as shared decision making between the physician and patient, recognizing both the personal motivation and the accountability on behalf of the patient (Hoskins et al. 2016).

This study aims to evaluate if the identification of a personalized outcome allows patients to achieve a better control of asthma in terms of asthma control test (ACT) and asthma quality of life questionnaire (AQLQ). In addition, a set of clinical outcomes (i.e. forced expiratory volume in one second - FEV1, use of rescue therapy, night awakeness) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥18 years;
2. Patients with a documented diagnosis of mild/moderate asthma, according to GINA, for at least 6 months before visit 1;
3. Patients on LABA/ICS chronic inhaled treatment (> 4 weeks before visit 1);
4. ACT values <20 points
5. No smoking patients, or former smokers (at least 1 year since quitting smoking, and no more than 10 pack/year, according the WHO definition);
6. Patients able to set up a personal outcome according to the protocol instruction, and willing to improve their personal outcome;
7. Patients able to understand written and spoken Italian;
8. Patients who give their informed consent to participate in the study.

Exclusion Criteria:

1. Patients treated with oral corticosteroids (OCS) and/or biological for severe refractory asthma;
2. Patients treated with OCS for any other chronic disease;
3. Subjects with current evidence of chronic obstructive pulmonary disease (COPD), pneumonia, active tuberculosis, active lung cancer, significant bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases or respiratory abnormalities other than asthma;
4. Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
5. Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome. The primary outcome of the study is to evaluate the impact of the personalized approach on asthma control (PDO group) versus a non-personalized approach (UC group). | Primary outcome will be measured at month 3 by asthma control test (ACT).
  The primary outcome of the study is to evaluate the impact of the personalized approach on asthma control (PDO group) versus a non-personalized approach (UC group). Primary outcome will be measured at month 3 by asthma control test (ACT).

SECONDARY OUTCOMES:
Secondary Outcome. To evaluate the impact of the personalized approach on asthma control (PDO group) versus a non-personalized approach (UC group) assessed by the change of ACT from month 3 to month 6. | from month 3 to month 6
  To evaluate the impact of the personalized approach on asthma control (PDO group) versus a non-personalized approach (UC group) assessed by the change of ACT from month 3 to month 6. Patients with an increase in the ACT score of 3 or greater will be considered responders. The secondary outcome will be calculated as the difference in percentage of the responders in each of the two groups;
Secondary outcome. To evaluate the impact of the personalized approach on asthma control (PDO group) versus a non-personalized approach (UC group) assessed by the change of AQLQ from baseline to month 3. | from baseline to month 3
  To evaluate the impact of the personalized approach on asthma control (PDO group) versus a non-personalized approach (UC group) assessed by the change of AQLQ from baseline to month 3. Patients with an increase in total AQLQ score of at least 0.5 points will be considered responders. The outcome will be calculated as the difference in percentage of the responders in each of the two groups.
Secondary outcome. To evaluate the impact of the personalized approach on asthma control (PDO group) versus a non-personalized approach (UC group) assessed by the change of AQLQ from month 3 to month 6. | from month 3 to month 6;
  To evaluate the impact of the personalized approach on asthma control (PDO group) versus a non-personalized approach (UC group) assessed by the change of AQLQ from month 3 to month 6. Patients with an increase in total AQLQ score of at least 0.5 points will be considered responders. The outcome will be calculated as the difference in percentage of the responders in each of the two groups.
Secondary outcome. To evaluate the impact of the personalized approach on asthma control assessed by the change of lung function (pulmonary functions tests: FEV1, FVC, FEV1/FVC) from baseline to month 3. | from baseline to month 3
  To evaluate the impact of the personalized approach on asthma control assessed by the change of lung function (pulmonary functions tests: FEV1, FVC, FEV1/FVC) from baseline to month 3.
Secondary outcome. To evaluate the impact of the personalized approach on asthma control assessed by the change of lung function (pulmonary functions tests: FEV1, FVC, FEV1/FVC) from baseline from month 3 to month 6. | from month 3 to month 6
  To evaluate the impact of the personalized approach on asthma control assessed by the change of lung function (pulmonary functions tests: FEV1, FVC, FEV1/FVC) from baseline from month 3 to month 6.
Secondary outcome. To measure the proportion of patients in the PDO group who achieve their own personal outcome at month 3, assessed by VAS (1-10) to V1. | at month 3
  To measure the proportion of patients in the PDO group who achieve their own personal outcome at month 3, assessed by VAS (1-10) to V1.
Secondary outcome. To measure the proportion of patients in the PDO group who achieve their own personal outcome at month 6, assessed by a VAS (1-10) as minimal clinically important difference (MCID) of 1.5 points to V1. | at month 6
  To measure the proportion of patients in the PDO group who achieve their own personal outcome at month 6, assessed by a VAS (1-10) as minimal clinically important difference (MCID) of 1.5 points to V1.
Secondary outcome. To measure the proportion of patients in the PDO group who maintain/improve their own personal outcome at month 6, assessed by a VAS (1-10) to V2. | at month 6
  To measure the proportion of patients in the PDO group who maintain/improve their own personal outcome at month 6, assessed by a VAS (1-10) to V2.

CONTACTS AND LOCATIONS:
Locations (12):
- Italy (12):
  - ASST Papa Giovanni XXIII, Bergamo
  - Azienda ospedaliera Spedali Civili di Brescia, Brescia
  - Ospedale San Martino di Genova, Genova
  - ASST Fate Bene e Fratelli Sacco, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - ASST Santi Paolo e Carlo, Milan
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico Milano, Milan
  - Policlinico San Matteo, Pavia
  - Ospedale di Rovigo, Rovigo
  - Humanitas Hospital - UO Allergologia, Rozzano
  - Humanitas Hospital - UO Pneumologia, Rozzano
  - Istituti Clinici Scientifici Maugeri, IRCCS Tradate, Tradate

IPD SHARING:
Plan to Share IPD: Undecided